CLINICAL TRIAL: NCT00802230
Title: Beta-Receptor SELECTivity of Carvedilol and Metoprolol Succinnate in Patients With Heart Failure: A Randomized Dose Ranging Trial (SELECT Trial)
Brief Title: Pharmacodynamic Study of Carvedilol Versus Metoprolol in Heart Failure
Acronym: SELECT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Edward M. Gilbert, M.D.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Select-B1B2
Record Dates: First submitted 2008-12-02; First posted 2008-12-04 (Estimated); Last update posted 2023-11-08 (Actual); Status verified 2008-12

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Carvedilol IR
  Interventions: Drug: Terbutaline Infusion
- 2 (Active Comparator): Metoprolol Succinate
  Interventions: Drug: Terbutaline Infusion

INTERVENTIONS:
Drug: Terbutaline Infusion

SUMMARY:
Metoprolol succinate is a beta1-selective beta-blocker, becoming non-selective at higher doses, while carvedilol is non-selective. We examined whether metoprolol remained beta1-selective compared to carvedilol during dose up-titration in Class C heart failure (HF) Beta-blocker naïve patients.

METHODS: Twenty-five NYHA FC II-III HF patients were randomized to carvedilol or metoprolol. Patients were studied at baseline and after 2 weeks of up-titration (metoprolol at 25, 50, 100, and 200 mg daily; carvedilol IR at 3.125, 6.25, 12.5, 25 mg and 50mg twice daily). Beta2- blockade was determined by an infusion of terbutaline at 6 mg/kg over 1 hour. Glucose and potassium levels were serially measured at baseline, every 15 minutes for the 1st hour and 30 minutes for 2nd hour post-infusion. The median area under the curve (AUC) for glucose and potassium changes were calculated.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for the study had objective evidence of systolic dysfunction (ejection fraction ≤40%), were >18 years of age, and were on stable optimal medical heart failure therapy excluding the use of beta-blockers within the previous 30 days.

Exclusion Criteria:

* . Patients were excluded for active viral myocarditis; hemodynamically significant valvular heart disease; hypertrophic cardiomyopathy, peripartum cardiomyopathy; contra-indications to beta-blockers (asthma or obstructive airway disease requiring scheduled bronchodilators or inhaled steroids), resting heart rate <55; supine blood pressure <85/50; second or third degree heart block); concomitant use of beta-agonists, beta-antagonists, or anti-arrhythmics; unstable angina; myocardial infarction or bypass surgery within 3 months; or significant renal insufficiency (creatinine >2.5 mg/dL), liver disease (transaminase levels > 3 fold above laboratory normal), or anemia.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2002-09; Primary Completion 2004-12 (Actual); Study Completion 2004-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Utah, Salt Lake City, Utah, United States